CLINICAL TRIAL: NCT05604989
Title: Associations Between the Oral and Intestinal Microbiome and Neovascular Age-related Macular Degeneration and the Investigation on the Effect of Oral Probiotics as a Treatment - A Pilot Study
Brief Title: Associations Between the Oral and Intestinal Microbiome and Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, KWANGSIC JOO, Director, Deparment of Ophthalmology, Principal Investigator, Clinical Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AMDMICROBIOME
Record Dates: First submitted 2022-10-17; First posted 2022-11-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-12

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: neovascular AMD; microbiome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neovascular AMD patients with anti-VEGF treatment, oral probiotics supplement (Experimental): Neovascular AMD patients will be allocated. Regular intravitreal anti-VEGF injection treatment will be done. At the baseline and 6 months, the investigators will collect stool, saliva, and blood samples for microbiome analysis.
  Oral probiotics (The Perfect Probiotics®) supplement will be given to the participants for 6 months.
  Interventions: Drug: Probiotic Combination Cap/Tab; Drug: intravitreal Anti-VEGF injection
- neovascular AMD patients with anti-VEGF treatment, no oral probiotics supplement (Sham Comparator): Neovascular AMD patients will be allocated. Regular intravitreal anti-VEGF injection treatment will be done. At the baseline and 6 months, the investigators will collect stool, saliva, and blood samples for microbiome analysis.
  No Oral probiotics (The Perfect Probiotics®) supplement in this group.
  Interventions: Drug: intravitreal Anti-VEGF injection
- Control patients, no oral probiotics supplement (No Intervention): Healthy, no retinal disease patients will be allocated. At the baseline and 6 months, the investigators will collect stool, saliva, and blood samples for microbiome analysis.
  No Oral probiotics (The Perfect Probiotics®) supplement in this group.

INTERVENTIONS:
Drug: Probiotic Combination Cap/Tab — The Perfect Probiotics® capsule will be given as an intervention, which is composed of mostly Lactobacillus acidophilus & Bifidobacterium lactis.
  Other Names: The Perfect Probiotics®
  Arms: Neovascular AMD patients with anti-VEGF treatment, oral probiotics supplement
Drug: intravitreal Anti-VEGF injection — Intravitreal anti-VEGF injection treatment in the neovascular AMD patients.
  Arms: Neovascular AMD patients with anti-VEGF treatment, oral probiotics supplement; neovascular AMD patients with anti-VEGF treatment, no oral probiotics supplement

SUMMARY:
A pilot study for Associations between the oral and intestinal microbiome and neovascular age-related macular degeneration and the investigation on the effect of oral probiotics as a treatment

The investigators recruit the neovascular AMD patients and control patients.

1. 15 neovascular AMD patients with anti-VEGF treatment and oral probiotics supplement
2. 15 neovascular AMD patients with anti-VEGF treatment and no oral probiotics supplement
3. 15 control patients and no oral probiotics supplement

The investigators will collect stool, blood, and saliva sample at the baseline and 6 months, and analyze the oral and intestinal microbiome changes.

ELIGIBILITY:
Inclusion Criteria:

* Normal BMI patients
* Diagnosed as neovascular AMD (experimental & sham group)
* Normal patients (control group)

Exclusion Criteria:

* Obese (BMI > 30)
* Past surgical history involving intestinal diseases
* Previous oral antibiotic treatment before 1 week at the baseline enroll
* Previous oral probiotics supplement
* Previous ophthalmic retinal diseases except neovascular AMD

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Oral microbiome changes after oral probiotics supplement in neovascular AMD patients | 6 months after enrollment
  The investigators will analyze the oral microbiome changes (baseline and 6 months after taking oral probiotics) in experimental, sham, and control groups.
  Microbiome relative abundance changes in percentage (%) will be statistically analyzed between baseline and 6 months.
Intestinal microbiome changes after oral probiotics supplement in neovascular AMD patients | 6 months after enrollment
  The investigators will analyze the intestinal microbiome changes (baseline and 6 months after taking oral probiotics) in experimental, sham, and control groups.
  Microbiome relative abundance changes in percentage (%) will be statistically analyzed between baseline and 6 months.

SECONDARY OUTCOMES:
Visual acuity changes after oral probiotics supplement | 6 months after enrollment
  If possible, visual acuity difference between experimental and sham group (oral probiotics vs. no oral probiotics) in the neovascular AMD patients.
  Visual acuity will be measured by the ETDRS eye chart (scale : letters).

CONTACTS AND LOCATIONS:
Overall Officials: Kwangsic Joo, MD PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No